CLINICAL TRIAL: NCT05033639
Title: Efficacy Of Oral Melatonin To Prevent Necrotizing Enterocolitis Among Preterm Infants In A Tertiary Level Hospital In The Philippines: A Randomized Control Trial
Brief Title: Efficacy Of Oral Melatonin To Prevent Necrotizing Enterocolitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ilocos Training and Regional Medical Center (Other Government)
Collaborators: Vayu Global Foundation (Unknown)
Responsible Party: Principal Investigator, Navid Roodaki, Pediatric Chief Resident, Ilocos Training and Regional Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ITRMC-REC-2021-008
Record Dates: First submitted 2021-08-22; First posted 2021-09-05 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Necrotizing Enterocolitis
MeSH Terms: conditions — Enterocolitis, Necrotizing | interventions — Melatonin; Milk, Human

STUDY DESIGN:
Intervention Model Description: This is a double-blind Randomized Control trial where melatonin would be the interventions given to preterm infants admitted at the Neonatal Intensive Care Unit of Ilocos Training and Regional Medical Center.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Once the mother is admitted for labor, she or the father will be asked to sign consent. However, if the mother was admitted as an emergency delivery, the parents would be ask immediately after delivery. No one would know what group the patient will be. Enrolled infants will be randomized by a 1:1 block scheme to provide a comparable subject in each group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Other than the Standard Management of preterm infant, treatment group A infants will receive 6 mg tablet dissolved in 5 ml breastmilk via oral gastric tube administered once a day at 10 pm.
  Interventions: Drug: Melatonin 6 MG
- Control Group (Placebo Comparator): Human breast milk 5ml would be used as the placebo in this study. It would be indistinguishable from the treatment group as this will also be the diluent used.
  Interventions: Other: Breast Milk

INTERVENTIONS:
Drug: Melatonin 6 MG — Melatonin is an endogenously produced indolamine principally synthesized in the pineal gland from serotonin. It is described as a ubiquitous molecule which plays a vital role in the physiologic function of the body. Melatonin, also known as N-acetyl-5-methoxytryptamine which has a a) immunomodulator; b) free radical scavenger; c) prevention of oxidative stress and d) anti-inflammatory7-10.
  Arms: Treatment Group
Other: Breast Milk — Naturally occurring milk from the mother of the infant.
  Arms: Control Group

SUMMARY:
Prematurity is still one of the primary causes of death in children under 5. 1-2. According to the WHO, 60% of all preterm births occur in Asia, with the Philippines accounting for around 348,900 every year. 3. Necrotizing enterocolitis is one of the fatal complications (NEC) 3, 4. Preterm newborns weighing 1500 grams or less are considered high risk. 5-6.

Melatonin is one chemical that may help prevent NEC. Melatonin is an endogenous indolamine derived from serotonin. It is a ubiquitous molecule that is crucial to the body's physiologic function. Melatonin, also known as N-acetyl-5-methoxytryptamine, is an immunomodulator, antioxidant, anti-inflammatory, and free radical scavenger7-10.

It is a naturally occurring chemical that is simply replenished. With this in mind, the researcher wants to see if providing high dose melatonin to premature babies can prevent NEC.

DETAILED DESCRIPTION:
Prematurity remains as one of the leading causes of mortality among children less than 5 years old1-2. The World Health Organization that 60 percent of all preterm births around the world occurs in Asian countries and roughly 348,900 births occur each year in the Philippines3. One complication that contribute to the high mortality is necrotizing enterocolitis (NEC)1, 3-4. High risk population include preterm infants weighing 1500 grams and lower with inverse correlation to the patient's weight5-6.

One compound that could be used to prevent NEC is melatonin. Melatonin is an endogenously produced indolamine principally synthesized in the pineal gland from serotonin. It is described as a ubiquitous molecule which plays a vital role in the physiologic function of the body. Melatonin, also known as N-acetyl-5-methoxytryptamine which has a a) immunomodulator; b) free radical scavenger; c) prevention of oxidative stress and d) anti-inflammatory7-10.

It is a naturally occurring substance and it would just be supplemented to increase its levels. With all this in mind, the researcher would like to determine if giving high dose melatonin among preterm neonates could prevent NEC among high risk population.

ELIGIBILITY:
Inclusion Criteria:

* 1. Newborn with a pediatric age of less than 37 weeks categorized very preterm (28 to 32 weeks) and late preterm (32 to 36weeks) by the World Health Organization weighing not more than 1500.

  2. Preterm infants admitted at the Neonatal Intensive care unit of Ilocos Training Regional and Medical Center not more than 24 hours of age.

  3. Preterm infants with orogastric tube in place. 4. Preterm infants with no other condition other than prematurity and respiratory distress syndrome.

  5. Preterm infant with an Apgar score of more than 6 in the first minute of life.

Exclusion Criteria:

1. Preterm infants more than 1 day of life.
2. Preterm infants diagnosed with NEC
3. Preterm infants who is born to a mother of who considered as a minor (<18 years old) and is not married to the father of the unborn child.
4. Preterm infants that could not be fed through oral gastric tube due to a secondary problem.
5. Preterm infants with other comorbidities such as asphyxia, congenital anomalies, and other inherited disorders.
6. Meconium Stained Preterm infants

   -

Ages: 28 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Number Of Preterm Infants Who Developed Necrotizing Enterocolits After Melatonin 6mg Tablet Prophylaxis | 5 MONTHS
  effectiveness of melatonin in preventing NEC among preterm infants with a birthweight of </ = 1500 kg at Ilocos Training and Regional Medical Center.

SECONDARY OUTCOMES:
Incidence of Prematurity at Training and Regional Medical Center | 5 MONTHS
  Clinical Profiles Of Preterm Infants Born In Ilocos Training and Regional Medical Center
Number of Patients Who Developed Abnormal Gas Pattern with Dilated Bowel Loops after Melatonin 6mg Tablet Prophylaxis | 5 MONTHS
  Absence of Clinical And Radiologic Findings Diagnostic of Necrotizing Enterocolitis.
Number of Patients Who Developed Pneumatosis intestinalis after Melatonin 6mg Tablet Prophylaxis | 5 Months
  Absence of Clinical And Radiologic Findings Diagnostic of Necrotizing Enterocolitis.
Number of Patients Who Developed Sentinel Loops after Melatonin 6mg Tablet Prophylaxis | 5 Months
  Absence of Clinical And Radiologic Findings Diagnostic of Necrotizing Enterocolitis.
Number of Patients Who Developed Portal Venous Gas after Melatonin 6mg Tablet Prophylaxis | 5 Months
  Absence of Clinical And Radiologic Findings Diagnostic of Necrotizing Enterocolitis.
Number Of Hospital Days Among Preterm Infants Admitted at Ilocos Training and Regional Medical Center | 5 Months
  Efficacy of Melatonin Oral Prophylaxis
Number Of Days Before Oral FeedingAmong Preterm Infants Admitted at Ilocos Training and Regional Medical Center | 5 motnhs
  Efficacy of Melatonin Oral Prophylaxis

CONTACTS AND LOCATIONS:
Overall Officials: Daisy Evangeline C Garcia, MD, Study Director — Ilocos Training and Regional Medical Center; Navid P Roodaki, MD, Principal Investigator — ITRMC
Locations (1):
- Ilocos Training and Regional Medical Center, San Fernando City, LA Union, Philippines

IPD SHARING:
Plan to Share IPD: No
due to the data privacy act of the philippines, individual data cannot be shared however the completed data will be shared